CLINICAL TRIAL: NCT02203656
Title: Feasibility Study of Post-hospitalization Interventions to Improve Physical Function
Brief Title: Feasibility Study of Post-hospitalization Interventions to Improve Physical Function in Older Adults
Acronym: PACE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Dairy Research Institute (Other); National Dairy Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 13-038; 1229 (Other Grant/Funding Number: Dairy Research Institute)
Record Dates: First submitted 2014-05-22; First posted 2014-07-30 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2017-12

CONDITIONS: Aging
Keywords: intervention studies; nutrition; exercise; testosterone; patient readmission
MeSH Terms: conditions — Motor Activity | interventions — Dietary Supplements; Testosterone; testosterone enanthate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo Supplement (Placebo Comparator): Daily placebo supplement for 30 days after discharge.
  Interventions: Drug: Placebo
- Nutritional Supplement (Experimental): Daily nutritional supplement for 30 days after discharge.
  Interventions: Dietary Supplement: Nutritional Supplement
- In-home exercise + placebo (Experimental): in-home exercise 3 times a week and daily placebo supplement for 30 days after discharge.
  Interventions: Drug: Placebo; Behavioral: In-home exercise
- In-home exercise + nutrition (Experimental): in-home exercise 3 times a week and daily nutritional supplement for 30 days after discharge.
  Interventions: Dietary Supplement: Nutritional Supplement; Behavioral: In-home exercise
- Testosterone (Experimental): Single testosterone injection within 24 hours of hospital discharge.
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Placebo — placebo supplement
  Other Names: Control
  Arms: In-home exercise + placebo; Placebo Supplement
Dietary Supplement: Nutritional Supplement — protein supplement
  Arms: In-home exercise + nutrition; Nutritional Supplement
Behavioral: In-home exercise — In-home exercise program
  Arms: In-home exercise + nutrition; In-home exercise + placebo
Drug: Testosterone — Testosterone injection
  Other Names: Testosterone enanthate
  Arms: Testosterone

SUMMARY:
The purpose of this study is to test the feasibility of interventions to accelerate recovery of muscle mass and function in older adults following acute hospitalization.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility of interventions to accelerate recovery of muscle mass and function in older adults following acute hospitalization

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the University of Texas Medical Branch (UTMB) ACE unit with an admitting diagnosis of congestive heart failure, respiratory infection, kidney/urinary tract infection, or metabolic disorder; or other condition that will allow a subject to participate in the study after patient review
* Aged 65 years or older
* Self-reported ability (with or without the aid of an assistive device) to walk across a small room two weeks prior to hospitalization
* Lives within 30 miles of UTMB
* Can stand without assistance at the time of pretesting
* Presents no medical contraindication to wearing a loose fitting velcro strap for the accelerometer on one ankle
* Score ≥26 on the 30-item Mini Mental State Examination or alert and oriented X3 by physician on H&P
* Is discharged "to home" at ACE unit discharge.

Exclusion Criteria:

* Nursing home resident or hospice patient
* Uncontrolled blood pressure (systolic >150, or diastolic > 100)
* History of stroke with motor disability
* Glomerular filtration rate (GFR) <30 mL/min/1.73m2 or evidence of kidney disease or failure
* Liver disease ( aspartate aminotransferase (AST) /Alanine transaminase (ALT) 2 times above the normal limit, hyperbilirubinemia)
* Recent (within 3 months) treatment with anabolic steroids
* Any other condition or event considered exclusionary by the PI and faculty physician
* Planned or elective hospitalization within 30 days of discharge

Additional Exclusion Criteria for Subjects Randomized to the Testosterone Group

* Breast or prostate cancer
* Palpable prostate nodule or induration or prostate specific antigen (PSA) ≥ 4 ng/ml
* PSA ≥ 3 ng/ml in men at high risk of prostate cancer, such as African Americans or men with first-degree relatives with prostate cancer
* Hematocrit ≥ 50%
* Decompensated heart failure as determined by a physician

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 113 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery- Gait, Balance, Chair Rise changes in functional measure score | at pre-testing, 1-week post discharge and 4-week post discharge
  Changes in SPPB score

SECONDARY OUTCOMES:
Body Composition | at pre-testing, 1-week post discharge and 4-week post discharge
  Body composition will be measured using a bioimpedance scale. Changes in weight and % body fat will be calculated over the duration of the intervention.
Hand grip strength (kg) | at pre-testing, 1-week post discharge and 4-week post discharge
  Changes in hand grip will be calculated over duration of study.
ADLS, IADLS | at pre-testing, 1-week post discharge and 4-week post discharge
  Changes in Instrumental activities of daily living (IADLS), and Activities of daily living (ADLS) will be measured over the duration of the intervention.
Physical Activity Levels | at pre-testing, 1-week post discharge and 4-week post discharge
  Physical activity levels will be measured using a step activity monitor and actiwatch
Gait Speed (m/s) | at pre-testing, 1-week post discharge and 4-week post discharge
  Changes in gait speed will be calculated over duration of study.
Blood Measures | at pre-testing, 1-week post discharge and 4-week post discharge
  microRNA levels in blood will be measured
30 day re-hospitalization | 30 days post-discharge
  re-hospitalization rates will be collected

OTHER OUTCOMES:
Follow-up Measures | 1 year post discharge
  Rehospitalization: date of rehospitalization, duration, and discharge diagnosis Death: date of death

CONTACTS AND LOCATIONS:
Overall Officials: Elena Volpi, MD, PhD, Principal Investigator — UTMB
Locations (2):
- United States (2):
  - UTMB Acute Care for Elders Unit, Galveston, Texas
  - Jennie Sealy Hospital, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No
No. This is a small Phase 1 pre-pilot study. Risk of loss of confidentiality

REFERENCES:
- [Background] Deer RR, Dickinson JM, Fisher SR, Ju H, Volpi E. Identifying effective and feasible interventions to accelerate functional recovery from hospitalization in older adults: A randomized controlled pilot trial. Contemp Clin Trials. 2016 Jul;49:6-14. doi: 10.1016/j.cct.2016.05.001. Epub 2016 May 10. PMID 27178766
- [Result] Deer RR, Goodlett SM, Fisher SR, Baillargeon J, Dickinson JM, Raji M, Volpi E. A Randomized Controlled Pilot Trial of Interventions to Improve Functional Recovery After Hospitalization in Older Adults: Feasibility and Adherence. J Gerontol A Biol Sci Med Sci. 2018 Jan 16;73(2):187-193. doi: 10.1093/gerona/glx111. PMID 28591764
- [Result] Deer RR, Dickinson JM, Baillargeon J, Fisher SR, Raji M, Volpi E. A Phase I Randomized Clinical Trial of Evidence-Based, Pragmatic Interventions to Improve Functional Recovery After Hospitalization in Geriatric Patients. J Gerontol A Biol Sci Med Sci. 2019 Sep 15;74(10):1628-1636. doi: 10.1093/gerona/glz084. PMID 30906944
- [Derived] Arentson-Lantz EJ, Deer RR, Kokonda M, Wen CL, Pecha TA, Carreon SA, Ngyen TM, Volpi E, Nowakowski S. Improvements in sleep quality and fatigue are associated with improvements in functional recovery following hospitalization in older adults. Front Sleep. 2022;1:1011930. doi: 10.3389/frsle.2022.1011930. Epub 2022 Oct 14. PMID 37251511